CLINICAL TRIAL: NCT01687296
Title: A Multicentre, Randomized, Double-blind, Double-dummy, Active-controlled, Parallel-group Study to Determine the Efficacy and Safety of Nebulized Fluticasone Propionate 1mg Twice Daily Compared With Oral Prednisone Administered for 7 Days to Chinese Pediatric and Adolescent Subjects (Aged 4 to 16 Years) With an Acute Exacerbation of Asthma
Brief Title: Nebulized Fluticasone Propionate VS Oral Prednisone in Chinese Pediatric and Adolescent Subjects With an Acute Exacerbation of Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114220
Record Dates: First submitted 2012-09-06; First posted 2012-09-18 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: PEF; inhaled; Fluticasone Propionate; safety; prednisone; acute exacerbation; asthma; efficacy
MeSH Terms: conditions — Asthma; Respiratory Aspiration | interventions — Prednisone; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluticasone Nebules/placebo tablet (Experimental): 2×0.5mg/2ml twice daily neblulized/placebo tablet, oral, once daily
  Interventions: Drug: fluticasone propionate inhalation solution; Drug: placebo tablet; Drug: salbutamol
- oral prednisone/placebo inhalation solution (Active Comparator): once daily (2mg/kg.day, up to 40mg/day for 4 days, then 1mg/kg.day or half of the original dose, up to 20mg/day for 3 days) / placebo inhalation solution nebulized twice daily
  Interventions: Drug: oral prednisone; Drug: placebo inhalation solution; Drug: salbutamol

INTERVENTIONS:
Drug: fluticasone propionate inhalation solution — 2×0.5mg/2ml twice daily nebulized to treat an acute exacerbation of asthma for 7 days
  Arms: fluticasone Nebules/placebo tablet
Drug: oral prednisone — once daily (2mg/kg.day, up to 40mg/day for 4 days, then 1mg/kg.day or half of the original dose, up to 20mg/day for 3 days) to treat an acute exacerbation of asthma for 7 days
  Arms: oral prednisone/placebo inhalation solution
Drug: placebo inhalation solution — 4ml 0.9% saline nebulized twice daily
  Arms: oral prednisone/placebo inhalation solution
Drug: placebo tablet — placebo soluble tablet, oral ,once daily
  Arms: fluticasone Nebules/placebo tablet
Drug: salbutamol — Salbutamol MDI 2 puffs twice daily or Nebules twice daily, and can be increased up to every 4 hours on an as-needed basis, through the treatment period.

SUMMARY:
This is a multicentre, randomized, double-blind, double-dummy, active-controlled, parallel-group study to determine the efficacy and safety of nebulized fluticasone propionate 1mg twice daily compared with oral prednisone administered for 7 days to Chinese pediatric and adolescent subjects (aged 4 to 16 years) with an acute exacerbation of asthma

DETAILED DESCRIPTION:
This is a multicentre, randomized, double-blind, double-dummy, active-controlled, parallel-group study to determine the efficacy and safety of nebulized fluticasone propionate (FP) 1mg twice daily compared with oral prednisone administered for 7 days to Chinese pediatric and adolescent subjects (aged 4 to 16 years) with an acute exacerbation of asthma. This study is for supporting registration of FP Nebules treating Chinese pediatric and adolescent subjects (aged 4 to 16 years) with an acute exacerbation of asthma in China.

At least 250 subjects, aged 4-16 years old, diagnosed an acute exacerbation of asthma at presentation, are eligible to take part in the study if they meet the inclusion criteria. They are randomly assigned at the ratio 1:1 to one of the following treatment groups for 7 days: FP Nebules 2×0.5mg/2ml twice daily/Placebo tablets once daily; Or, Oral prednisone tablets once daily (2mg/kg.day, up to 40mg/day for 4 days, then 1mg/kg.day or half of the original dose, up to 20mg/day for 3 days) / Placebo Nebules 2×2ml 0.9% saline twice daily. While all subjects are given Salbutamol Nebules / MDI for relief of symptoms. After randomization (visit 1), the following visits are on Day5 (visit 2) and Day8 (visit 3), and a follow-up phone call (visit4) will happen two weeks post treatment on Day 21 for collection of adverse events.

The primary endpoint is mean morning PEF on diary card over the treatment assessment period. The secondary endpoints include subject derived data (symptom scores ), evening PEF on diary card, use of rescue medications, clinic assessments of pulmonary function ( FEV1, and FVC) , clinical scoring index , patient/parent and investigator global evaluation, and use of rescue medications during the trial. Safety endpoints include AEs, vital signs, and oropharyngeal examinations, and laboratory tests (haematology, urinalysis, chemistry). The subjects are assessed for compliance on completion of diary card.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male and female pediatric or adolescent subjects aged 4 to 16 years, inclusive
* Subjects have an established diagnosis of asthma
* The definition of asthma. According to Chinese Guideline for the diagnosis and optimal management of asthma in children [Respiratory branch of pediatric society,Chinese Medical. Association. 2008, revised version], the subjects can be diagnosed when meeting the criteria. The diagnosis criteria is listed in the protocol.
* The severity of an acute exacerbation of asthma is defined as PEF of 50% to 75% predicted via a peak flow meter, with a clinical scoring index of ≥2. The clinical scoring index represents the sum of the score for each of four signs: respiratory rate (0=low to 3=high, dependent on age), wheezing (0=none to 3=severe), inspiration/expiration ratio (0=2:1 to 3=1:3), and accessory muscle (0=none to 3=marked use).
* Subjects can properly use a mini-wright peak flow meter, nebulizer and MDI with/without a spacer, and accurately complete a diary card with parental assistance, if required.
* Subjects' parents/guardians are willing to give written informed consent.

Exclusion criteria:

* Severe respiratory dysfunction.
* History of mechanical ventilation due to respiratory failure.
* Admission to hospital due to respiratory disease within the previous 2 weeks, including asthmatic exacerbations.
* Clinical or lab evidence of a serious, uncontrolled systemic disease or presence of any disease likely to interfere with the objectives of this study, such as pulmonary cystic fibrosis and bronchopulmonary dysplasia.
* Known or suspected hypersensitivity to glucocorticosteroids or β2 agonists.
* Clinical visual evidence of oral candidiasis at Visit1.
* Use of the medications below in Table 1 according to the following defined time intervals prior to presentation. The list is provided in the protocol.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 261 (Actual)
Dates: Start 2012-11-12; Primary Completion 2013-06-01 (Actual); Study Completion 2013-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- China (9):
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Yanji, Jilin
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Wenzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Wuxi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned on 250 Chinese paediatric and adolescent participants (aged 4 to 16 years) with an acute exacerbation of asthma and was conducted at 11 centres in China from 12th November 2012 to 21st June 2013.
Pre-assignment Details: A total of 266 participants (par) were screened for this study. Of these, 5 participants were screen failures. A total of 261 participants were randomized to receive either nebulized fluticasone or oral prednisone. A total of 251 participants received at least a single dose study drug.
Groups:
- Fluticasone Propionate: Participants received fluticasone propionate inhalation solution twice daily (BID) 2x0.5 milligrams (mg)/millilitres (mL) via a nebulizer in morning and evening for 7 days. Blinding was maintained by administration of placebo soluble tablets once daily in the morning for 7 days. Salbutamol was provided on a needed basis throughout the treatment period.
- Prednisone: Participants received oral prednisone tablets once daily at 2 mg per kilogram (kg) per day, up to 40 mg per day for 4 days, then 1 mg per kg per day or half of the original dose, up to 20 mg per day for 3 days in the morning. Blinding was maintained by administration of placebo nebules 2×2mL 0.9% saline BID in morning and evening for 7 days. Salbutamol was provided on a needed basis throughout the treatment period.
Period: Overall Study
Arm/Group | Fluticasone Propionate | Prednisone
Started | 123 | 128
Completed | 116 | 123
Not Completed | 7 | 5
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Fluticasone Propionate: Participants received fluticasone propionate inhalation solution BID 2x0.5 mg/mL via a nebulizer in morning and evening for 7 days. Blinding was maintained by administration of placebo soluble tablets once daily in the morning for 7 days. Salbutamol was provided on a needed basis throughout the treatment period.
- Prednisone: Participants received oral prednisone tablets once daily at 2 mg per kg per day, up to 40 mg per day for 4 days, then 1 mg per kg per day or half of the original dose, up to 20 mg per day for 3 days in the morning. Blinding was maintained by administration of placebo nebules 2×2mL 0.9% saline BID in morning and evening for 7 days. Salbutamol was provided on a needed basis throughout the treatment period.
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate | Prednisone | Total
Number analyzed (Participants) | 123 | 128 | 251
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.6 (2.41) | 6.5 (2.32) | 6.5 (2.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 51 | 102
  Male | 72 | 77 | 149
Region of Enrollment [Number; unit: Participants]
  China | 123 | 128 | 251

OUTCOME MEASURES:

1. Primary Outcome: Mean Morning Peak Expiratory Flow (AM PEF) on Diary Card Over the Treatment Assessment Period in Intent-to-Treat (ITT) Population
Description: PEF is the maximum flow generated during a forceful exhalation, starting from full lung inflation. Participants (if needed with the help of parents or guardian) recorded on diary card the best of three PEF measurements, using a mini-Wright peak flow meter in the morning before taking any study drug. Only data that was drawn from Days 2 to 8 after randomization and on or before one day after the end date of study drug was used for analysis. The outcome measure was considered missing if less than 2 days were recorded in the given treatment assessment period. Two participants from fluticasone propionate group and 4 participants from prednisone group had the missing outcome measure. Analysis was performed using an analysis of covariance (ANCOVA) model with effects due to gender, age, centre and treatment group.
Time Frame: Days 2 to 8
Population: ITT Population comprised of all participants randomized to treatment and who received at least one dose of study drug. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Litres per minute (L/min)
Arm/Group | Fluticasone Propionate | Prednisone
Number analyzed (Participants) | 121 | 124
Litres per minute (L/min) | 188.77 (3.774) | 188.31 (3.790)
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Prednisone; 250 par were to be enrolled to achieve 200 total evaluable par or 100 evaluable par per group. Sample size was based on the primary efficacy endpoint (AM PEF) and had 80% power to reject the null hypothesis: nebulized FP (1 mg BID) was inferior to oral prednisone with regard to AM PEF using one-side t test at significance level 2.5%, and assuming true treatment difference (FP minus predisone) was 3.6 L/min, noninferiority margin was -12L/min, and common standard deviation was 39 L/min; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated at the lower limit of the 95% confidence interval (5%, 2-sided significance level) for the treatment difference (FP minus prednisone) in the mean morning PEF on diary card over the treatment assessment period was greater than -12L/min; p = 0.931, ANCOVA; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-9.85 to 10.76]

2. Primary Outcome: Mean Morning PEF on Diary Card Over the Treatment Assessment Period in Per Protocol (PP) Population
Description: PEF is the maximum flow generated during a forceful exhalation, starting from full lung inflation. Participants (if needed with the help of parents or guardian) recorded on diary card the best of three PEF measurements, using a mini-Wright peak flow meter in the morning before talking any study drug. Only data that was drawn from Days 2 to 8 after randomization and on or before one day after the end date of study drug was used for analysis. The outcome measure was considered missing if less than 2 days were recorded in the given treatment assessment period. Two participants from fluticasone propionate group and 5 participants from prednisone group had the missing outcome measure. Analysis was performed using ANCOVA model with effects due to gender, age ,centre and treatment group.
Time Frame: Days 2 to 8
Population: PP Population comprised of all participants in the ITT Population who did not have any full protocol violations which could impact treatment effect. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Fluticasone Propionate | Prednisone
Number analyzed (Participants) | 114 | 120
L/min | 189.46 (3.724) | 188.96 (3.712)
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Prednisone; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.922, ANCOVA; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-9.64 to 10.65]

3. Secondary Outcome: Mean Evening PEF on Diary Card Over the Treatment Assessment Period
Description: PEF is the maximum flow generated during a forceful exhalation, starting from full lung inflation. Participants recorded on diary card the best of three PEF measurements, using a mini-Wright peak flow meter in the evening (6:00-9:00 post meridiem [PM]) before taking any study drug. Only data that was drawn from Days 1/2 to 8 after randomization and before or on the end date of study drug was used for analysis. If participants started to take the study drug in the morning (early or on 12:00 PM), only then the evening PEF on the date of randomization was used. The outcome measure was considered missing if less than 2 days was recorded in the given treatment assessment period. Two participants from fluticasone propionate group and 5 participants from prednisone group had the missing outcome measure. Analysis was performed using an ANCOVA model with effects due to gender, age, centre and treatment group.
Time Frame: Days 1/2 to 8
Population: ITT Population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Fluticasone Propionate | Prednisone
Number analyzed (Participants) | 121 | 123
L/min | 195.79 (3.723) | 194.63 (3.751)
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Prednisone; Test type: Superiority or Other; p = 0.822, ANCOVA; Mean Difference (Final Values) = 1.16, 95% CI 2-sided [-9.02 to 11.34]

4. Secondary Outcome: Median Day-time and Night-time Symptom Scores Over the Treatment Assessment Period
Description: The symptoms of cough, sputum production, wheeze and dyspnoea were assessed in morning and evening, and recorded on participant diary cards. Day-time symptoms were scored while retiring to bed on a scale of 0 (no symptoms) to 5 (severe). Night-time symptoms were scored while waking in the morning on a scale of 0 (no symptoms) to 4 (severe). For day-time score, only data that was from Days 2 to 8 after randomization and before or on the end date of study drug was used. For night-time score, only data that are from Days 2 to 8 after randomization and on or before one day after the end date of study drug was used. The outcome measure was considered missing if less than 2 days were recorded in the given treatment assessment period. The analysis only includes participants with at least 2 days of non-missing symptom scores in the given treatment assessment period.
Time Frame: Days 2 to 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Fluticasone Propionate | Prednisone
Number analyzed (Participants) | 123 | 128
Scores on a scale
  Day-time symptom score: number analyzed (Participants) | 121 | 123
  Day-time symptom score | 0.5 [0 to 3] | 1.0 [0 to 3]
  Night-time symptom score: number analyzed (Participants) | 121 | 124
  Night-time symptom score | 0.0 [0 to 3] | 0.0 [0 to 4]
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Prednisone; Fluticasone propionate versus Prednisone for day-time symptom score; Test type: Superiority or Other; p = 0.717, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Fluticasone Propionate vs Prednisone; Fluticasone propionate versus Prednisone for night-time symptom score; Test type: Superiority or Other; p = 0.683, Wilcoxon rank sum test

5. Secondary Outcome: Median Number of Use of Rescue Medications During Day and Night Over the Treatment Assessment Period
Description: The use of nebulized salbutamol (doses/puffs and frequency) were recorded on diary card in the morning and evening. The median numbers of times of use of rescue medication during day and night was calculated for each participant over the treatment assessment period. In each case, only data that was from Days 2 to 8 after randomization and before or on the end date of study drug was used. The outcome measure was considered missing if less than 2 days (that is., 24-hour periods) were recorded in the given treatment assessment period. The analysis only includes participants who have at least 2 days of non-missing numbers of times rescue medication (including zero) in the given treatment assessment period.
Time Frame: Days 2 to 8
Population: ITT Population. Data is presented for the participants available at the time of assessment.
Measure: Median (Full Range); unit: Number of use of rescue medication
Arm/Group | Fluticasone Propionate | Prednisone
Number analyzed (Participants) | 121 | 123
Number of use of rescue medication | 2.0 [0 to 3] | 2.0 [0 to 3]
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Prednisone; Test type: Superiority or Other; p = 0.996, Wilcoxon rank sum test

6. Secondary Outcome: Clinical Assessment of Lung Function of Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC) During the Treatment Period
Description: Spirometric assessments of FEV1 and FVC were assessed at clinic visit 1 (Screening), 2 (Day 5) and 3 (Day 8). Lung function tests were performed at the approximately same time at each visit in the morning. Participants were instructed to withhold salbutamol therapy for at least 4 hour, and the highest of three FEV1 and FVC measurements were recorded. If participants discontinued before or on Day 5, then the FEV1 and FVC collected at the early withdrawal visit is included in the Visit 2. Otherwise, the FEV1, FVC collected at the early withdrawal visit was included in the Visit 3. Analysis was performed using ANCOVA with covariates of gender, centre, age and treatment.
Time Frame: During the treatment period at Day 5, Day 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Fluticasone Propionate | Prednisone
Number analyzed (Participants) | 123 | 128
Litres
  FEV1, Day 5: number analyzed (Participants) | 102 | 114
  FEV1, Day 5 | 1.288 (0.0348) | 1.331 (0.0332)
  FEV1, Day 8: number analyzed (Participants) | 103 | 118
  FEV1, Day 8 | 1.400 (0.0294) | 1.396 (0.0280)
  FVC, Day 5: number analyzed (Participants) | 107 | 118
  FVC, Day 5 | 1.476 (0.0454) | 1.543 (0.0439)
  FVC, Day 8: number analyzed (Participants) | 109 | 121
  FVC, Day 8 | 1.544 (0.0326) | 1.582 (0.0316)
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Prednisone; Fluticasone propionate versus Prednisone for FEV1 on Day 5; Test type: Superiority or Other; p = 0.348, ANCOVA; Mean Difference (Final Values) = -0.044, 95% CI 2-sided [-0.135 to 0.048]
Statistical Analysis 2: Comparison: Fluticasone Propionate vs Prednisone; Fluticasone propionate versus Prednisone for FEV1 on Day 8; Test type: Superiority or Other; p = 0.914, ANCOVA; Mean Difference (Final Values) = 0.004, 95% CI 2-sided [-0.074 to 0.083]
Statistical Analysis 3: Comparison: Fluticasone Propionate vs Prednisone; Fluticasone propionate versus Prednisone for FVC on Day 5; Test type: Superiority or Other; p = 0.276, ANCOVA; Mean Difference (Final Values) = -0.067, 95% CI 2-sided [-0.187 to 0.054]
Statistical Analysis 4: Comparison: Fluticasone Propionate vs Prednisone; Fluticasone propionate versus Prednisone for FVC on Day 8; Test type: Superiority or Other; p = 0.384, ANCOVA; Mean Difference (Final Values) = -0.039, 95% CI 2-sided [-0.126 to 0.049]

7. Secondary Outcome: Mean Change From Baseline in Clinical Scoring Index at Day 5 and Day 8
Description: The clinical scoring index was assessed at Baseline (Visit 1), Day 5 and Day 8. The score assigned represented the sum of the score for each of four signs: respiratory rate, wheezing, inspiration/expiration ratio, and accessory muscle use. Each of these parameters were scored on a 4-point scale of 0 to 3 where 0=none, 1=mild, 2=moderate and 3=severe. The total score ranged from 0 to 12, where 0 indicated absence of symptoms and 12 indicated most severe symptoms. The Baseline value was the last non-missing value prior to randomization. Change from Baseline was calculated/defined as value at the indicated visit minus value at the Baseline. A negative value of change in score from Baseline indicated improvement in severity of symptoms. If participants discontinued before or on Day 5, then the clinical scoring index collected at the early withdrawal visit was included in the Visit 2. Otherwise, the clinical scoring index collected at the early withdrawal visit was included in the Visit 3
Time Frame: Baseline, Day 5 and Day 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Fluticasone Propionate | Prednisone
Number analyzed (Participants) | 123 | 128
Scores on a scale
  Day 5: number analyzed (Participants) | 121 | 125
  Day 5 | -2.7 (1.41) | -2.6 (1.44)
  Day 8: number analyzed (Participants) | 116 | 123
  Day 8 | -3.4 (1.26) | -3.4 (1.26)
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Prednisone; Fluticasone propionate versus Prednisone for clinical scoring index on Day 5; Test type: Superiority or Other; p = 0.507, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Fluticasone Propionate vs Prednisone; Fluticasone propionate versus Prednisone for clinical scoring index on Day 8; Test type: Superiority or Other; p = 0.700, Wilcoxon rank sum test

8. Secondary Outcome: Mean Global Evaluation for Efficacy by Participant/Parent and Investigator
Description: At Visit 3 (Day 8), participant/parent and investigator were asked to evaluate efficacy globally as very beneficial=1, beneficial=2, no effect=3 or worse=4. The global evaluation collected at the early withdrawal visit was included in the Visit 3. If participants were discontinued at Visit 2, then the global evaluation collected at the Visit 2 is also included in the Visit 3 for summary and analysis.
Time Frame: Day 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Fluticasone Propionate | Prednisone
Number analyzed (Participants) | 123 | 128
Scores on a scale
  Participant/parent global evaluation: number analyzed (Participants) | 122 | 128
  Participant/parent global evaluation | 1.5 (0.59) | 1.5 (0.52)
  Investigator global evaluation: number analyzed (Participants) | 121 | 128
  Investigator global evaluation | 1.5 (0.56) | 1.5 (0.52)
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Prednisone; Fluticasone propionate versus Prednisone for participant/parent global evaluation; Test type: Superiority or Other; p = 0.633, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Fluticasone Propionate vs Prednisone; Fluticasone propionate versus Prednisone for investigator global evaluation; Test type: Superiority or Other; p = 0.323, Wilcoxon rank sum test

ADVERSE EVENTS:
Time Frame: On- treatment serious adverse events (SAE) and non- serious adverse events (AE) were collected from start of study medication through the treatment phase up to 8 days (only on-treatment events captured).
Description: Safety Population comprised of participants randomized to treatment and who receive d at least one dose of study drug. Participants were assigned to the treatment group as per treatment actually received.
Arm/Group | Fluticasone Propionate | Prednisone
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/128
Serious Adverse Events (participants affected / at risk) | 1/123 | 2/128
Other Adverse Events (participants affected / at risk) | 1/123 | 10/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Propionate (N=123) | Prednisone (N=128)
Upper respiratory tract infection (Infections and infestations) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Propionate (N=123) | Prednisone (N=128)
White blood cell count increased (Investigations) | 1 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.